CLINICAL TRIAL: NCT06172972
Title: Atraumatic Care Practice From the Child and Parent Perspective
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Hatice Uzşen, Principal Investigator, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Atraumatic Care
Record Dates: First submitted 2023-11-27; First posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Nurse's Role
Keywords: child; fear; pain; phlebotomy; distraction methods; atraumatic care
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atraumatic nursing care group (Experimental): Before the phlebotomy, children in the intervention group were allowed to choose a distracting method (foam balloons, stress balls, musical books) to be occupied with during the procedure. It was ensured that the parent was staying with the child and that the child played with this material during the procedure (making a foam balloon, squeezing the ball with the hand in which the procedure was not carried out and reading the book with the parent
  Interventions: Behavioral: Atraumatic nursing care
- Control group (No Intervention): The parents of the children in the control group were ensured to stay with their children during the procedure, and the child's attention was distracted by the nurse asking questions about the child's name, age, and what grade the child was in. This is one of the methods frequently used in Turkiye.

INTERVENTIONS:
Behavioral: Atraumatic nursing care — Children in the intervention group were allowed to choose a distracting method (foam balloons, stress balls, musical books) to be occupied with during the procedure
  Arms: Atraumatic nursing care group

SUMMARY:
It is important for pediatric nurses to apply atraumatic care while providing care to children and their families. Pediatric nurses should use methods appropriate for the child's age and developmental period within the scope of atraumatic care.

DETAILED DESCRIPTION:
The use of atraumatic care approaches such as supporting the active participation of the family in the care of the child, using therapeutic communication techniques with parents and children during procedures, providing emotional support, reducing pain during painful procedures, using techniques to distract the child's attention during medical procedures, informing parents about the procedures to be performed on their children, and supporting parents and teaching techniques to cope with stress is recommended to be used by the nurses.

ELIGIBILITY:
Inclusion Criteria:

* being able to speak Turkish
* being between 5-10 years of age
* having no visual, intellectual or neurological disabilities
* having the phlebotomy procedure carried out with a single attempt
* not having a disease that causes chronic pain
* being accompanied by either mother or father during the procedure
* not taking painkillers or sedating drugs before the phlebotomy procedure

Exclusion Criteria:

* being younger than 5 years or older than 10 years
* having visual, audio, or speech impairments
* having a disease that causes chronic pain
* with a history of sedative and analgesic use within 24 h prior to admission
* filling out the data collection forms incompletely

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 219 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Children's Fear Scale | baseline, pre-intervention and immediately after the intervention
  Children's Fear Scale was to measure fear in children who would undergo painful medical procedures
Wong-Baker Faces Pain Rating Scale | immediately after the intervention
  This scale is used for 3-18 age group children to describe their pain.

SECONDARY OUTCOMES:
Assessment of Parental Satisfaction-Visual Analog Scale | immediately after the intervention
  Parent satisfaction scores were collected using a question about care satisfaction during the phlebotomy procedure from each child's parent.

CONTACTS AND LOCATIONS:
Overall Officials: Esra Tural Büyük, PhD, Study Chair — Ondokuz Mayıs University
Locations (1):
- Hatice Uzşen, Samsun, Atakum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.